CLINICAL TRIAL: NCT01728038
Title: Exploring a Cessation Intervention for Low Income Smokers in an Emergency Setting
Brief Title: Exploring a Cessation Intervention for Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIN381902; 1K22CA163747 (NIH)
Record Dates: First submitted 2012-11-13; First posted 2012-11-16 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: Bronchiolitis; Cough; Ear Infection; Respiratory Infection; Wheezing
MeSH Terms: conditions — Asthma; Bronchiolitis; Cough; Otitis; Respiratory Tract Infections; Respiratory Sounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cessation Counseling (Experimental): Parental smokers will be given a brief cessation intervention consisting of counseling, nicotine replacement therapy and Quitline connection.
  Interventions: Behavioral: Cessation Counseling

INTERVENTIONS:
Behavioral: Cessation Counseling — Parental Smokers will be given brief cessation counseling, nicotine replacement therapy and Quitline connection.

SUMMARY:
An estimated 6.6 million parents who smoke visit pediatric emergency departments (PED) annually. Up to 50% of these parental smokers are from low-income, racially/ethnically diverse households in which a variety of tobacco-related disparities (TRD) exist for both the parents and their children. The PED is an ideal setting in which to address these disparities, which include differences in tobacco use, pediatric second hand smoke exposure (SHSe), quit rates, access to cessation resources, and morbidity such as cancer. The team has conducted the only two small-scale randomized control trials (RCTs) investigating the efficacy of providing smoking cessation counseling to parents in the PED setting. This previous research indicates that parental smokers who visit the PED are aware of the pediatric effects of SHSe, motivated to quit, eager to receive cessation counseling in this setting, and show trends towards quitting.

Parents with children who have a SHSe-related illness will have higher prolonged abstinence and point prevalence cessation rates, higher motivation to quit, greater number of quit attempts, and lower child SHSe compared to those parents who have a child with a non-SHSe-related illness at baseline.

DETAILED DESCRIPTION:
The long-range goal of my research is to test PED-based cessation interventions that are readily translated into practice in large, multi-center trials. However, before this can occur, preliminary data are needed, including analyses of: (1) the types of cessation intervention components that low-income parental smokers regard as essential to their cessation success; (2) perceived organizational barriers to the sustainability of the intervention after the study period ends which will impede translation into practice; (3) factors associated with parental cessation outcomes such as the presence of an acute SHSe-related chief complaint in the child; and (4) the effect size of the intervention. This data will be used to develop a parental cessation intervention that is tailored to low-income parents who are likely to quit. Data from the proposed project will be used in a RO1 application to test the efficacy of this cessation intervention in a large, multi-center randomized trial.

The proposed developmental study will be conducted in three phases. During Phase I, the investigators will conduct focused interviews of PED nurses, physicians, and hospital administrators to explore barriers to intervention sustainability that will assist in future intervention planning. During Phase II, The investigators will conduct a pilot prospective trial to examine the effectiveness of this screening, brief intervention, and assisted referral to treatment (SBIRT) intervention on parental smoking cessation. Equal numbers of parental smokers who bring their child to the PED for either a SHSe-related illness or non SHSe-related illness will be given a brief intervention using an adapted form of the Clinical Practice Guidelines: Treating Tobacco Use and Dependence. Intervention components may include brief cessation counseling using an "Advise, Assess, and Assist" approach; information on SHSe in children; direct connection to the Quitline (QL) in the ED; and/or free administration of nicotine replacement therapy (NRT). The Health Belief Model will be used to explore whether factors unique to this setting (e.g., child's acute illness) moderate the effect of the intervention on cessation outcomes. Outcomes will be assessed following the intervention via phone, email, or text messaging, based on parental preference. In Phase III we will explore the feasibility of a pilot study to collect, send, analyze, and store child saliva samples in twenty five children whose parents consent to the study. The same PED-based SBIRT cessation intervention will be given to these parental smokers as in Specific Aim 2, however, only English-speaking parents and parents of children who are 0-5 years of age who present to the PED with SHSe-related illnesses will be asked if they agree to have their child participate in this baseline and then 1-month after baseline, saliva sample collection. These saliva samples will be analyzed to assess child cotinine levels at baseline and again at 1 month after the SBIRT cessation intervention. Leftover saliva will be stored and frozen indefinitely for possible future research, if parents consent.

ELIGIBILITY:
Phase 1: Focused Interviews of Pediatric Emergency Department Practitioners will be conducted to assess their perceived attitudes and barriers to implementing routine tobacco screening and tobacco counseling in the pediatric emergency department.

Inclusion Criteria:

* Hospital personnel: PED medical director, Chief of Staff, Chairman of Pediatrics, quality systems specialists, informational technology specialists, PED physicians, and PED registered nurses.

Exclusion Criteria:

* Non-hospital personnel

Phase 2: Parental smokers who bring their children to the pediatric emergency department will be given brief smoking cessation counseling which includes advice on quitting, nicotine replacement therapy vouchers and direct Quitline connection.

Inclusion Criteria:

* Parent/Legal Guardian (18 years or older), who are tobacco users, accompanying a child (0 to 18 years old) being treated in the PED with a non-urgent complaint/condition.

Exclusion Criteria:

* Parent/Legal Guardian who is only a tobacco chewer.
* Parent/Legal Guardian who is enrolled in a smoking cessation program.
* Parent/Legal Guardian who is using Nicotine Replacement Therapy (NRT) or other cessation treatment.
* Parent/Legal Guardian who is moving within 8 months after enrollment.

Phase 3: The same PED-based SBIRT cessation intervention will be given to these parental smokers as in Phase 2. However, parents will also be asked if they agree to have their child participate in saliva sample collection at baseline and at one month. Parents will also be asked if their child's leftover saliva can be stored for future research.

Inclusion Criteria:

* Parent/Legal Guardian (18 years or older), who are tobacco users, accompanying a child (0 to 5 years old) being treated in the PED with a non-urgent second hand smoke exposure related complaint/condition.

Exclusion Criteria:

* Parent/Legal Guardian who is only a tobacco chewer.
* Parent/Legal Guardian who is enrolled in a smoking cessation program.
* Parent/Legal Guardian who is using Nicotine Replacement Therapy (NRT) or other cessation treatment.
* Parent/Legal Guardian who is moving within 8 months after enrollment
* Parent/Legal Guardian who does not speak or read English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Parents who report that they have not smoked in the past seven (7) days, and their verbal response is verified by a carbon monoxide test. | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Esther M. Mahabee-Gittens, MD, MS, Principal Investigator — Professor
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Mahabee-Gittens EM, Stone L, Gordon JS. Pediatric emergency department is a promising venue for adult tobacco cessation interventions. Nicotine Tob Res. 2013 Oct;15(10):1792-3. doi: 10.1093/ntr/ntt069. Epub 2013 May 24. No abstract available. PMID 23709612
- [Result] Mahabee-Gittens EM, Khoury JC, Ho M, Stone L, Gordon JS. A smoking cessation intervention for low-income smokers in the ED. Am J Emerg Med. 2015 Aug;33(8):1056-61. doi: 10.1016/j.ajem.2015.04.058. Epub 2015 May 2. PMID 25976268